CLINICAL TRIAL: NCT06371456
Title: Anon Invasive Confirmatory Sign for Correct Epidural Catheter Placement During Normal Vaginal Delivery
Brief Title: A Non Invasive Confirmatory Sign for Correct Epidural Catheter Placement During Normal Vaginal Delivery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ain Shams university 111
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Normal Delivery Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- epidural anesthesia (Experimental)
  Interventions: Procedure: epidural catheter placement

INTERVENTIONS:
Procedure: epidural catheter placement — after sterilization of the back, local anesthesia injection (xylocaine 5 ml) at lumbar 4-5 level, then advancing the epidural needle till loss of resistance by air occurs and the epidural catheter inserted then aspiration through the catheter will be done to confirm that no accidental cerebrospinal fluid or blood are aspirated and to observe the dew sign inside the outer portion of the epidural catheter near the back of the patient

SUMMARY:
Epidural anesthesia for pain control during normal vaginal delivery is a blind maneuver and so we need a confirmatory sign for being in the correct epidural space.

Loss of resistance sign using air may guide us wrongly as it may occur if we entered into the paravertebral muscles or cavities in the interspinal ligaments.

So, additional confirmatory sign beside loss of resistance sign by air is strongly needed.

We noticed that after occurence of loss of resistance sign by air and insertion of the epidural catheter a dew was formed on the internal sides of the epidural catheter after aspiration to be sure that there are no blood or cerebrospinal fluid in the catheter.

This dew formation (Ramy sign) is characteristic for air in the epidural space when transferred from the warm epidural space (temperature about 38-39 celsius degree) to the colder aspect of the catheter outside the patient which nearly has the same operating room temperature (22 celsius degree).

This sign may be associated with correct placement and good function of the epidural catheter.

DETAILED DESCRIPTION:
parturient for normal vaginal delivery are examined for correct epidural catheter placement by loss of resistance technique by air, observation of the dew sign and epidurogram.

Visual analogue score is used to test pain. blood pressure and heart rate after epidural injection will be monitored

ELIGIBILITY:
Inclusion Criteria:

* Parturient for normal vaginal delivery
* American society of anesthesiologists 2

Exclusion Criteria:

* patients refusal
* back infection
* anticoagulant non stopped
* platelets count less than 100000
* international normalization ratio more than 1.4
* severe cardiac or respiratory diseases
* haemodynamics unstable patients

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
appearance of the dew sign | immediately during aspiration of the epidural catheter
  dew formation inside the outer portion of the epidural catheter near the patient

SECONDARY OUTCOMES:
epidurogram | immediately after epidural catheter insertion
  by using posteroanterior x-ray image after injection of radiopaque dye through the epidural catheter with appearance of distribution of the dye in the epidural space and may exit through the neuroforamina laterally
visual analogue score | 20 minutes after epidural injection by 10 milliliter bupivacaine 0.25%
  making a handwritten mark on a 10 cm line that represents a continuum between "no pain" and "worst pain"
mean blood pressure | 20 minutes after epidural injection by 10 milliliter bupivacaine 0.25%
  by non invasive monitor
mean blood pressure | 30 minutes after epidural injection by 10 milliliter bupivacaine 0.25%
  by non invasive monitor
heart rate | 20 minutes after epidural injection by 10 milliliter bupivacaine 0.25%
  by non invasive monitor
heart rate | 30 minutes after epidural injection by 10 milliliter bupivacaine 0.25%
  by non invasive monitor